CLINICAL TRIAL: NCT00004421
Title: Phase II/III Study of Deep Brain Stimulation in Patients With Dystonia
Brief Title: Deep Brain Stimulation in Treating Patients With Dystonia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13315; MTS-FDR001452
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-03

CONDITIONS: Dystonia
Keywords: dystonia; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Dystonia; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Device: implanted pulse generator

SUMMARY:
RATIONALE: Dystonia is a disorder in which the muscles that control voluntary movements are persistently or intermittently contracted (not relaxed). Deep brain stimulation is provided by a small, battery operated implant placed under the skin of the chest that delivers low voltage electrical pulses through a wire under the skin that is connected to a specific area of the brain. Deep brain stimulation may help lessen the symptoms of dystonia.

PURPOSE: Phase II/III trial to study the effectiveness of deep brain stimulation in treating patients who have dystonia.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients undergo surgery to implant a brain stimulation system consisting of an implanted pulse generator (IPG) in the chest and a wire lead in the globus pallidum internal. After the lead has been implanted, the brain stimulation system is tested. Patients are examined at 1, 3, 6, 9, and 12 months after surgery. A double blinded evaluation, during which the IPG is either off or on, is carried out at 3 and 6 months.

Patients are followed every 3 months as long as the brain stimulation system remains in place.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Idiopathic or secondary cervical, segmental, or generalized dystonia not adequately controlled with traditional pharmacotherapy and/or botulinum toxin --Prior/Concurrent Therapy-- All medical therapy must be stable within the past month Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: No prior destructive neurosurgical procedure Other: At least 3 months since prior botulinum toxin injections --Patient Characteristics-- Age: 18 to 75 Performance status: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Cardiovascular: No demand cardiac pacemaker Other: No history of substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 1997-09; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Francis Brin, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, NY, New York, New York, United States

REFERENCES:
- [Background] Brin MF, Germano I, Danisi FO, et al.: Deep brain stimulation (DBS) of pallidum in intractable dystonia. Movement Disorders 13(suppl 2): 274, 1998.
- [Background] Germano IM, Villalobos H, Weisz, et al.: Image-guided computer-assisted technology as adjuvant for placement of deep brain stimulators. Movement Disorders 13(suppl 2): 264, 1998.